CLINICAL TRIAL: NCT04925999
Title: Distance Learning and Neck Disability Among Academic Staff During COVID-19 Period
Brief Title: Distance Learning and Neck Problems During Pandemic Period
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Misr University for Science and Technology (Other)
Responsible Party: Principal Investigator, Samah Mahmoud Sheha, principal investigator, Misr University for Science and Technology
Other Study IDs: P.T.REC/012/003211
Record Dates: First submitted 2021-06-08; First posted 2021-06-14 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Neck Pain
Keywords: Online Learning; Neck Pain; COVID-19
MeSH Terms: conditions — Neck Pain; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
For people who use computers a lot, Work-related musculoskeletal disorders of the neck are a common problem . It is generally agreed that the etiology of work-related neck disorders is multidimensional which is associated with, and influenced by, a complex array of individual, physical and psychosocial factors.

DETAILED DESCRIPTION:
Academic staff work involves diverse activities, both in and out of lecture-rooms, designing course curricula, developing lecture and tutorial plans and materials, providing students with information in an interesting and understandable manner, setting questions, and marking examinations .These activities usually involve long periods of sitting and standing, placing a physical demand on the lower back, cervical spine and the vertebral column in general, thus contributing to neck and shoulder discomfort .Lecturers use computers extensively and are thus exposed to many of the same risk factors to which 'office workers' are exposed. Using a computer is associated with poor neck posture most often in a forward head position, which is thought to be one of the most common causes of neck, head and shoulder tension and pain .

Neck pain is costly in terms of treatment, individual suffering, and time lost due to work absenteeism . Effective performance of academic staff of the university is very important as the key factors to a successful day to day running of any university system .

ELIGIBILITY:
Inclusion Criteria:

* At least one year of work experience in the current position as academic stuff.

Exclusion Criteria:

* Spinal deformities or specific medical condition affecting the cervical spine (e.g., ankylosing spondylitis, radiculopathy, tumors, infection and disc prolapse)
* History of spinal surgery
* Previous head or neck trauma

Ages: 25 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: * Both male and female working as academic staff at Misr University for Science and Technology.
  * Age range between 25 to 60 years old
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-06-15 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Neck disability index | 3 months
  It is designed to provide information as to how neck pain affects a person's ability to manage in everyday life

SECONDARY OUTCOMES:
Pain severity | 3 months
  Pain severity will be assessed using an 11- point numerical rating scale , where zero = no pain, 10 = unbearable pain. Each participant will rate the pain perceived along the scale at the point which refers to pain severity.

CONTACTS AND LOCATIONS:
Locations (1):
- Misr university for science and technology, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fejer R, Kyvik KO, Hartvigsen J. The prevalence of neck pain in the world population: a systematic critical review of the literature. Eur Spine J. 2006 Jun;15(6):834-48. doi: 10.1007/s00586-004-0864-4. Epub 2005 Jul 6. PMID 15999284
- [Background] Chiu TT, Lam PK. The prevalence of and risk factors for neck pain and upper limb pain among secondary school teachers in Hong Kong. J Occup Rehabil. 2007 Mar;17(1):19-32. doi: 10.1007/s10926-006-9046-z. PMID 16933144